CLINICAL TRIAL: NCT06788262
Title: Cerebral and Cognitive Modifications in Retired Female Professional Soccer Players as Compared to Non Exposed to Repeated Cranial Impacts Sportswomen : Transverse Analytic Study
Brief Title: Cerebral and Cognitive Impact of Female Professional SoccerPractice
Acronym: TCFOOT F
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 9414
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Chronic Encephalopathy
Keywords: soccer; MRI; head traumatism; neuropsychology; traumatic chronic encephalopathy
MeSH Terms: conditions — Chronic Traumatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Female professional Soccer players (Experimental): Diagnostic Test: MRI
  The following sequences of the MRI will be acquired during the inclusion visit:
  * 3D T1 gradient echo (GRE): anatomy; registration; cerebral, white matter, and grey matter volumetry; and cortical thickness;
  * multiecho 3D T2 GRE: quantitative susceptibility mapping (QSM), iron overload quantification;
  * continuous arterial spin labeling (ASL) 3D: cerebral perfusion;
  * resting-state fMRI: functional connectivity; -64-direction DTI (b=1000 and 2500): alterations in white matter and its microstructure, anatomic connectivity;
  * monovoxel spectroscopy of the mesencephalus with short echo time (TE).
  Interventions: Other: Cerebral MRI
- Female athletes not exposed to head injuries. (Active Comparator): Diagnostic Test: MRI
  The following sequences of the MRI will be acquired during the inclusion visit:
  * 3D T1 gradient echo (GRE): anatomy; registration; cerebral, white matter, and grey matter volumetry; and cortical thickness;
  * multiecho 3D T2 GRE: quantitative susceptibility mapping (QSM), iron overload quantification;
  * continuous arterial spin labeling (ASL) 3D: cerebral perfusion;
  * resting-state fMRI: functional connectivity;
  * 64-direction DTI (b=1000 and 2500): alterations in white matter and its microstructure, anatomic connectivity;
  * monovoxel spectroscopy of the mesencephalus with short echo time (TE).
  Interventions: Other: Cerebral MRI

INTERVENTIONS:
Other: Cerebral MRI — Cerebral MRI

SUMMARY:
The objective of this study is to evaluate, using MRI, the microstructural consequences and the onset of any cognitive impairment in female professional soccer players at the end of their career, who have experienced repeated minor head injuries. Over the long term, these head injuries could lead to morphological lesions and have an impact on female soccer players' cognitive skills.

The main evaluation criterion corresponds to the modifications found on MRI in the female professional soccer player group (diffusion tensor, cerebral perfusion, fMRI, cerebral volumetry and cortical thickness, spectroscopy, susceptibility imaging).

This is an exposure/nonexposure study assessing the onset of MRI abnormalities (diffusion tensor, cerebral perfusion, fMRI, volumetry and cortical thickness, spectroscopy, susceptibility imaging) in female professional soccer players exposed to repeated mild head injuries, who are either at the end of their career or retired for approximately 10 years, compared to high-level athletes not exposed to head injuries.

ELIGIBILITY:
Inclusion Criteria:

* Exposed high-level athletes: female professional soccer players at the end of their career (32- years old) playing in France Ligue 1 or 2 exposed to repeated mild head injuries with no history of severe head injury or cerebral
* Female High-level athletes not exposed to repeated mild head injuries: control group paired for age with female professional soccer players, who have never regularly participated in sports exposing them to head injuries (notably rugby, basketball, handball, American football, hockey, combat sports, etc.) and who have no history of head injury, even mild. Female Professional tennis players or former players will be preferentially recruited.

Exclusion Criteria:

* Refusal to be informed of abnormalities on MRI
* Incapacity to give informed consent or under a legal protection order;
* History of cerebral concussion including the presence after head shock of one or more of the following signs or symptoms: a period of confusion or disorientation, a period of loss of consciousness of 30 minutes or less, post-traumatic amnesia not exceeding 24 hours
* History of severe head/brain injury;
* History of neurological or psychiatric disorder;
* Known cerebral abnormality diagnosed by an imaging exam (CT or MRI);
* History or regular or occasional consumption of drugs, unweaned active smoking or weaned for less than 1 year, excessive consumption of alcohol (> 20 g alcohol per day, evaluated with the formula "degree of alcohol × volume in cl × 8/1000"), weaned or not.
* Usage of medication targeting the central nervous system in the 2 weeks preceding inclusion in the study;
* Prior history of severe hypertension, diabetes, chronic heart disease, progressive or disabling disease;
* Contraindication to MRI (claustrophobia, implanted material not compatible with MRI, refusal to be informed of abnormality discovered on MRI)

Ages: 32 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Cerebral MRI Microstructural abnormalities | Day 1
  Abnormalities on MRI in professional soccer players exposed to repeated mild head injuries, potentially related to chronic traumatic encephalopathy, compared to high-level athletes who are not exposed to head injuries.
  This is a study assessing the relation between exposure to mild head injuries during soccer play in professional players and the onset of MRI and neuropsychological abnormalities. The main evaluation criterion corresponds to the quantitative MRI modifications (professional soccer player group compared with control group).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane KREMER, MD, Principal Investigator — HOPITAUX UNIVERSITAIRES DE STRASBOURG